CLINICAL TRIAL: NCT04232995
Title: Efficacy of Balance Training in Comparison to General Exercises Alone in Diabetic Neuropathy
Brief Title: Balance Training in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Rabeiya Tazeem, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RTazeem
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Neuropathy With Neurologic Complication
Keywords: Diabetes Mellitus type 2; Diabetic neuropathy; Rehabilitation; Balance exercises; Berg Balance Scale
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Balance training by 9 positions with 1 min hold, repeated twice
  1. Stand with feet together, eyes remain open
  2. Stand with together, eyes closed
  3. & 4) Tandem Standing with Right and Left in front alternately
  5) Forward Reaching 6) & 7) Single Leg Standing, with Right and Left foot alternately 8) & 9) Step up, with Right and Left foot alternately
  General Exercises for 25 min
  * Active Range of Motion Exercises and Foot Care Education-5 min
  * Treadmill- 15 min
  * Cycling -5 min
  No. Of Sessions 24, thrice a week for 8 weeks
  Interventions: Other: Balance Training; Other: General Exercises
- Control Group (Active Comparator): General Exercises for 25 min
  * Active Range of Motion Exercises and Foot Care Education-5 min
  * Treadmill- 15 min
  * Cycling -5 min
  No. Of Sessions 24, thrice a week for 8 weeks
  Interventions: Other: General Exercises

INTERVENTIONS:
Other: Balance Training — Balance enhancing exercises
  Arms: Experimental Group
Other: General Exercises — General Exercises

SUMMARY:
This study evaluates the efficacy of balance training in Diabetic Neuropathy. Control group will receive general exercises while Eperimental/ Interventional group will receive Balance exercises along with general exercises.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 30-60 years
* Diabetes type II patients diagnosed with peripheral neuropathy by medical doctor for at least 5 years
* Neuropathy present (on the basis of Michigan Neuropathy Screening Instrument
* Have balance impairment ( evaluation on Berg Balance Scale)

Exclusion Criteria:

* Neuropathy due to other medical conditions like Vitamin deficiency, Hypothyroidism, Auto-immune/ demyelinating diseases
* Foot ulcers
* Lower limb amputee
* Vestibular diseases
* Retinopathy
* Cardiac problems
* Hemiplegia/ Stroke

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline (Pre treatment)
  The Berg Balance Scale (BBS) is a 56-point scale that evaluates 14 tasks. Katherine Berg developed this test to assess the level of function and balance in various patient populations. Minimum score is 0 (means severe balance deficit) and Maximum score is 56 (means No balance deficit)
Berg Balance Scale | At 4th week of treatment
  The Berg Balance Scale (BBS) is a 56-point scale that evaluates 14 tasks. Katherine Berg developed this test to assess the level of function and balance in various patient populations. Minimum score is 0 (means severe balance deficit) and Maximum score is 56 (means No balance deficit)
Berg Balance Scale | At 8th week of treatment (Post treatment )
  The Berg Balance Scale (BBS) is a 56-point scale that evaluates 14 tasks. Katherine Berg developed this test to assess the level of function and balance in various patient populations. Minimum score is 0 (means severe balance deficit) and Maximum score is 56 (means No balance deficit)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Physical Medicine and Rehabilitation, Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No